CLINICAL TRIAL: NCT00066079
Title: Home Based Massage and Relaxation for Sickle Cell Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001078-01A1 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Pain; Sickle Cell Disease; Chronic Pain; Alternative Medicine/Therapy; Complementary Medicine; Massage Therapy; Relaxation Technique; Home-based Therapy
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: massage
Behavioral: relaxation

SUMMARY:
The purpose of this study is to compare the effects of in-home, family-administered massage and in-home relaxation training on measures of physical status and health care utilization in a sample of African American adolescents age 15 years and older and adults with chronic pain associated with sickle cell disease who have been randomly assigned to six sessions of either family-administered massage or progressive muscle relaxation training.

ELIGIBILITY:
Inclusion criteria:

* Medically diagnosed with sickle cell disease, including hemoglobin SS disease, hemoglobin SD disease, hemoglobin SC disease, or sickle-thalassemia
* Self-report of having experienced chronic pain related to sickle cell disease during the past 30 days.
* Availability of a family member or friend who agrees to be trained to administer massages if the participant is randomized to the massage arm of the study.

Exclusion Criteria:

* Sickle cell trait instead of sickle cell disease diagnosis.
* Diagnosis of disease in addition to sickle cell disease which requires regular use of pain medication. (Please note, regular use of pain medication for sickle cell pain is NOT an exclusion)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia D. Myers, PhD, LMT, Principal Investigator — The Moffitt Cancer Center
Locations (2):
- United States (2):
  - Los Angeles Orthopaedic Hospital - Vascular Medicine Program, Los Angeles, California
  - Moffitt Cancer Center and Research Institute, Tampa, Florida

REFERENCES:
- [Background] Shapiro BS, Dinges DF, Orne EC, Bauer N, Reilly LB, Whitehouse WG, Ohene-Frempong K, Orne MT. Home management of sickle cell-related pain in children and adolescents: natural history and impact on school attendance. Pain. 1995 Apr;61(1):139-144. doi: 10.1016/0304-3959(94)00164-A. PMID 7644237
- [Background] Elander J, Midence K. A review of evidence about factors affecting quality of pain management in sickle cell disease. Clin J Pain. 1996 Sep;12(3):180-93. doi: 10.1097/00002508-199609000-00006. PMID 8866159
- [Background] Zeltzer L, Dash J, Holland JP. Hypnotically induced pain control in sickle cell anemia. Pediatrics. 1979 Oct;64(4):533-6. PMID 492819
- [Background] Co LL, Schmitz TH, Havdala H, Reyes A, Westerman MP. Acupuncture: an evaluation in the painful crises of sickle cell anaemia. Pain. 1979 Oct;7(2):181-185. doi: 10.1016/0304-3959(79)90009-5. PMID 523174
- [Background] Thomas JE, Koshy M, Patterson L, Dorn L, Thomas K. Management of pain in sickle cell disease using biofeedback therapy: a preliminary study. Biofeedback Self Regul. 1984 Dec;9(4):413-20. doi: 10.1007/BF01000558. PMID 6399460
- [Background] Cozzi L, Tryon WW, Sedlacek K. The effectiveness of biofeedback-assisted relaxation in modifying sickle cell crises. Biofeedback Self Regul. 1987 Mar;12(1):51-61. doi: 10.1007/BF01000078. PMID 3663738
- [Background] Wang WC, George SL, Wilimas JA. Transcutaneous electrical nerve stimulation treatment of sickle cell pain crises. Acta Haematol. 1988;80(2):99-102. doi: 10.1159/000205612. PMID 3138879
- [Background] Gil KM, Wilson JJ, Edens JL, Webster DA, Abrams MA, Orringer E, Grant M, Clark WC, Janal MN. Effects of cognitive coping skills training on coping strategies and experimental pain sensitivity in African American adults with sickle cell disease. Health Psychol. 1996 Jan;15(1):3-10. doi: 10.1037//0278-6133.15.1.3. PMID 8788535
- [Background] Gil KM, Carson JW, Sedway JA, Porter LS, Schaeffer JJ, Orringer E. Follow-up of coping skills training in adults with sickle cell disease: analysis of daily pain and coping practice diaries. Health Psychol. 2000 Jan;19(1):85-90. doi: 10.1037//0278-6133.19.1.85. PMID 10711591
- [Background] Dinges DF, Whitehouse WG, Orne EC, Bloom PB, Carlin MM, Bauer NK, Gillen KA, Shapiro BS, Ohene-Frempong K, Dampier C, Orne MT. Self-hypnosis training as an adjunctive treatment in the management of pain associated with sickle cell disease. Int J Clin Exp Hypn. 1997 Oct;45(4):417-32. doi: 10.1080/00207149708416141. PMID 9308268
- [Background] Jacobson E. 1974. Progressive muscle relaxation. Chicago: University of Chicago Press, Midway Reprint.
- [Background] Field TM. Massage therapy effects. Am Psychol. 1998 Dec;53(12):1270-81. doi: 10.1037//0003-066x.53.12.1270. PMID 9872050
- [Background] Myers CD, Robinson ME, Guthrie TH, Jr, Lamp SP, Lottenberg R. Adjunctive approaches for sickle cell chronic pain. Alternative Health Practitioner 1999;5:203-212.36.
- [Background] Benjamin LJ, Dampier CD, Jacox AK, Odesina V, Phoenix D, Shapiro B, Strafford M, Treadwell M. Guideline for the management of acute and chronic pain in sickle-cell disease. APS Clinical Practice Guidelines Series, No. 1. 1999. Glenview, IL: American Pain Society.